CLINICAL TRIAL: NCT06461494
Title: Comparative Effect of Egoscue Versus Pilates Exercises on Pain, Range of Motion, Flexibility and Muscles Endurance in Patients With Mechanical Low Back Pain
Brief Title: Comparison of Egoscue Versus Pilates Exercises in Patient With Mechanical Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/ 0195 Ghazala
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain
Keywords: muscle endurance; pain; range of motion; muscle flexibility
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Pilates exercise (Active Comparator): Group A received the pilates exercise. It doesn't require any special equipment and can be done in any training center.
  Week 1: Leg slides, hip release, knee to chest, spinal rotation, single knee extension, cat stretch, neutral to imprint Week 2: Imprint table top position, ab prep, Imprint table top toe touching floor, imprint table top knee extensions, spine twist, Ab prep in table top position, bridging Week 3: Half roll back, pull up; pull up with leg extension, swimming exercise, single leg extension, leg circles, and single leg stretch Week 4: Bridging on the ball, spine stretch forward, single leg lift, double knee lifts, upward dog, and shell stretch Each exercise was performed for 5 times
  Interventions: Other: baseline treatment
- Group B: Egoscue exercise (Experimental): Static back and static back with breathing, abdominal contraction while in the static back position, abductor press, overhead extension, elbow curls on wall, static wall, upper spinal twist, pelvic tilts, supine groin progressive, and air bench Week 1: 3 times with 30 s hold time Week 2: 5 times with 30 s hold time Week 3: 15 times with 30 s hold time Week 4: 20 times with 30 s hold time
  Interventions: Other: baseline treatment

INTERVENTIONS:
Other: baseline treatment — hot pack will be applied for 10 minutes

SUMMARY:
Mechanical low back pain arises intrinsically from the spine, intervertebral disc,or surrounding soft tissues.It is causes by muscular spasm, and other soft tissue injuries. The aim of the study will be to compare the effect of Egoscue versus Pilates exercises on pain, range of motion and muscle endurance in patient with mechanical low back pain.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at Riphah Clinic Lahore through consecutive sampling technique on 30 patients which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with Pilates exercises at frequency 2 sets 5 repetitions 5 days a week and Group B will be treated with Egoscue exercises at the frequency of 2 sets with 5 repetitions 5 days a week. Outcome measures will be conducted through pain, disability,lumber range of motion, Muscle flexibility, Extensor muscle endurance, Lateral muscle endurance, Flexors muscle endurance questionnaires after 4 weeks. Data will be analyzed during SPSS software version 21. After assessing normality of data by ANOVA test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years
* Both gender
* Patient with non-radiating pain
* Pain NPRS <7
* Positive McGill Extensor Endurance Test ( <101 seconds)
* Positive McGill lateral flexor endurance test (<54 sec Right side, <55sec left side)
* Positive McGill flexor endurance test < 120 seconds
* Positive Finger to Floor Test : > 48cm in males, >50cm for females
* Patient with Oswestry disability index (ODI) < 40 ODI score
* Decrease lumbar ROM; Lateral flexion, Extension, Flexion

Exclusion Criteria:

* Sacroiliac Joint Dysfunction (SIJD)
* Coccydynia
* Lumber disc pathology
* Malignancy
* Recent fractures

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | upto 4 weeks
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Muscle flexibility (Finger to floor test) | upto 4 weeks
  * The patient is asked to bend forward and attempt to reach for the floor with their fingertips.
  * The physical therapist then measures the distance between the patient's right long finger and the floor using a standard measuring tape
  * Ask the client whether pain, stiffness or both limit the movement(Fingertips to floor (FTF) test).
  * If the FTF test is limited by pain, the location and pain score out of 10 should be documented.
  * If the FTF test is 0cm or the patient is able to place their palms to the floor with no pain, a different outcome measure should be considered.
Trunk Flexor Endurance Test | upto 4 weeks
  The flexor endurance test is the first in the battery of three tests that assesses muscular endurance of the deep core muscles (i.e., transverse abdominis, quadratus lumborum, and erector spinae). It is a timed test involving a static, isometric contraction of the anterior muscles, stabilizing the spine until the individual exhibits fatigue and can no longer hold the assumed position.
Trunk Lateral Endurance Test | upto 4 weeks
  The trunk lateral endurance test, also called the side-bridge test, assesses muscular endurance of the lateral core muscles (i.e., transverse abdominis, obliques, quadratus lumborum, and erector spinae). Similar to the trunk flexor endurance test, this timed test involves static, isometric contractions of the lateral muscles on each side of the trunk that stabilize the spine.
Trunk Extensor Endurance Test | upto 4 weeks
  The trunk extensor endurance test is generally used to assess muscular endurance of the torso extensor muscles (i.e., erector spinae, longissimus, iliocostalis, and multifidi). This is a timed test involving a static, isometric contraction of the trunk extensor muscles that stabilize the spine.
universal goniometer | upt0 4 weeks
  The purpose of goniometry is to measure the joint angle or range of motion. It is assumed that the angle created by aligning the arms of a universal goniometer with bony landmarks truly represents the angle created by the proximal and distal bones composing the joint.

CONTACTS AND LOCATIONS:
Overall Officials: Ghazala Arshad, MSPT*, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Med care hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kudchadkar GS, Gurudut P, Welling AJIJoPT, Research. Comparative effect of mat pilates and egoscue exercises in asymptomatic individuals with lumbar hyperlordosis: A randomized controlled trial. 2019;1(2):79-88.
- [Background] Baillie L, Bacon CJ, Hewitt CM, Moran RW. Predictors of functional improvement in people with chronic low back pain following a graded Pilates-based exercise programme. J Bodyw Mov Ther. 2019 Jan;23(1):211-218. doi: 10.1016/j.jbmt.2018.06.007. Epub 2018 Jun 30. PMID 30691755
- [Background] Altinbilek T, Murat S. A comparison of application frequency of physical therapy modalities in patients with chronic mechanical low back pain. Turk J Phys Med Rehabil. 2020 May 18;66(2):201-209. doi: 10.5606/tftrd.2020.4192. eCollection 2020 Jun. PMID 32760898
- [Background] Jerome EJIJoP. Effects of core stabilization program and conventional exercises in the management of patients with chronic mechanical low back pain. 2015:441-7.
- [Background] Caglayan M, Tacar O, Demirant A, Oktayoglu P, Karakoc M, Cetin A, et al. Effects of lumbosacral angles on development of low back pain. 2014;22(3):251-5.
- [Background] Kumar SP. Efficacy of segmental stabilization exercise for lumbar segmental instability in patients with mechanical low back pain: A randomized placebo controlled crossover study. N Am J Med Sci. 2011 Oct;3(10):456-61. doi: 10.4297/najms.2011.3456. PMID 22363083
- [Background] Russo M, Deckers K, Eldabe S, Kiesel K, Gilligan C, Vieceli J, Crosby P. Muscle Control and Non-specific Chronic Low Back Pain. Neuromodulation. 2018 Jan;21(1):1-9. doi: 10.1111/ner.12738. Epub 2017 Dec 12. PMID 29230905
- [Background] Vining R, Potocki E, Seidman M, Morgenthal AP. An evidence-based diagnostic classification system for low back pain. J Can Chiropr Assoc. 2013 Sep;57(3):189-204. PMID 23997245